CLINICAL TRIAL: NCT00415272
Title: Pulmonary Rehabilitation in Patients With Fibrotic Interstitial Lung Disease
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Inadequate enrollment.
Sponsor: University of California, San Francisco (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H52476-29802-01
Record Dates: First submitted 2006-12-20; First posted 2006-12-22 (Estimated); Last update posted 2008-01-15 (Estimated); Status verified 2008-01

CONDITIONS: Fibrotic Interstitial Lung Disease

INTERVENTIONS:
Behavioral: Pulmonary Rehabilitation

SUMMARY:
Our study aims to investigate the benefits of an outpatient pulmonary rehabilitation program in a population of subjects with fibrotic interstitial lung disease. Our hypothesis is that pulmonary rehabilitation will lead to improvements in quality of life, breathlessness, exercise capacity and pulmonary function in this patient population.

ELIGIBILITY:
Inclusion Criteria:

1. Restriction on pulmonary function testing (TLC <80%, FEV1/FVC ratio > predicted or DLCO < 80%)
2. Evidence of fibrosis on high resolution computed tomography of the chest.
3. Fibrosis on surgical lung biopsy if performed
4. Referral for pulmonary rehabilitation

Exclusion Criteria:

1. Participation in pulmonary rehabilitation in the past 24 months
2. Inability to complete 6 minute walk test or study questionnaires
3. Limitations other than dyspnea (e.g. arthritis) that affect ability to participate in pulmonary rehabilitation
4. Baseline 6 minute walk distance > 400 meters
5. Planned change in medication treatment for lung disease during the course of pulmonary rehabilitation
6. Ejection fraction known to be < 25%
7. Contraindications to pulmonary rehabilitation (clinically unstable, uncontrolled arrhythmia or hypertension, symptomatic or uncontrolled hypotension with systolic blood pressure of < 95, active angina, unexplained syncope or worsening dizziness, limiting orthopedic or neurological disorders, psychiatric impairment that inhibits cooperation in the program)
8. FEV1/FVC < 65%
9. Unable to provide informed consent

Sex: All
Age Groups: Child, Adult, Older Adult
Dates: Study Completion 2007-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Harold R Collard, MD, Principal Investigator — University of California at San Francisco
Locations (1):
- University of California at San Francisco, San Francisco, California, United States